CLINICAL TRIAL: NCT06525038
Title: PRISMA 7 (for Frailty Assessment) and SARC-F (for Evaluation of Sarcopenia Risk) in Predicting Emergency Department Readmission and Mortality
Brief Title: PRISMA 7 and SARC-F in Predicting Emergency Department Readmission and Mortality
Status: Completed | Type: Observational
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Mehmet Cagri Goktekin, Assoc. Prof., Firat University
Other Study IDs: FiratU-EM-MCG-01
Record Dates: First submitted 2024-07-19; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Frailty; Sarcopenia; Morality
Keywords: Emergency Service; Mortality; Sarcopenia; Frailty
MeSH Terms: conditions — Frailty; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Risk of sarcopenia (-) and risk of frailty (-)
  Interventions: Other: All groups were observed for clinical end-points described in the study protocol
- Risk of sarcopenia (+) and risk of frailty (-)
  Interventions: Other: All groups were observed for clinical end-points described in the study protocol
- Risk of sarcopenia (-) and risk of frailty (+)
  Interventions: Other: All groups were observed for clinical end-points described in the study protocol
- Risk of sarcopenia (+) and risk of frailty (+)
  Interventions: Other: All groups were observed for clinical end-points described in the study protocol

INTERVENTIONS:
Other: All groups were observed for clinical end-points described in the study protocol — All groups were observed for clinical end-points (mortality, readmission to emergency service) described in the study protocol.

SUMMARY:
Frailty scores can predict hospitalization and other related adversities. Thus, the frailty status determination is useful in clinical decisions regarding elderly patients. This study aimed to evaluate the potential of PRISMA-7 and SARC-F scores in predicting hospitalization following emergency department (ED) admission, readmission at 1, 3, and 6 months, and mortality within a 6-month follow-up period.

DETAILED DESCRIPTION:
1. Aim Most screening tools for frailty and sarcopenia are complex and thus impractical for emergency physicians. They require more time. Administering them to patients in limited time and in emergencies is difficult as it requires most equipment. Among these methods, PRISMA-7 and SARC-F can be applied in the ED as they are practical, fast, and convenient.

   This prospective study evaluates the ability of PRISMA-7 and SARC-F to predict hospitalization after ED admission, readmission to the hospital ED at 1, 3, and 6 months, and mortality at 6-month follow-up.
2. Materials and Methods 2.1 Study Design and Compliance Criteria This study was approved by the Non-Interventional Research Ethics Committee of Firat University and conducted by the Faculty of Medicine, Department of Emergency Medicine. 150 patients aged ≥65 who presented to the emergency department (ED) in a 6-month period from January 2023 to July 2023 were included in this study. The patient's gender, comorbidities, and reasons for admission were examined. The admission dates to the ED were recorded. Patients and their relatives were informed about the study to obtain written informed consent.

Patients meeting the inclusion criteria and providing written consent to participate in this study were included. The patients were consecutively included in the study. Patients with no spontaneous heartbeat or breathing at the time of ED arrival, the ones refusing to participate in the study, and whose information could not be retrieved were excluded. The patients' SARC-F and PRISMA-7 scores were calculated at the first ED presentation. Later, the same patients were evaluated via the electronic hospital system and called by phone. Their status was assessed regarding the recurrent ED visits, hospitalization, and mortality at 1, 3, and 6 months. Patients were divided into four groups. Group 1: risk of sarcopenia (-) and risk of frailty (-), Group 2: risk of sarcopenia (+) and risk of frailty (-), Group 3: risk of sarcopenia (-) and risk of frailty (+), and Group 4: risk of sarcopenia (+) and risk of frailty (+).

2.2 Frailty and Sarcopenia Assessment PRISMA-7 assessment included seven yes/no questions. The questionnaire interrogated patients' demographic characteristics (age and gender), physical ability, limiting medical problems, and dependency on others. The questionnaire was scored between 0 and 7 points, where higher scores indicated higher severity of frailty. A score of ≥3 suggested further assessment and that the patient had a frailty risk. Turkish validity and reliability studies of this questionnaire were conducted.

The SARC-F for sarcopenia assessment had five questions. Each question was scored between 0 and 2. The questionnaire interrogated patients' strength, assistance in walking, climbing stairs, rising from chairs, and falling status. The questionnaire was scored between 0 and 10 points. A score of ≥4 demonstrated possible sarcopenia risk and indicated the need for the patient's further examination. It was susceptible for detecting sarcopenia risk in older adults.

2.3 Follow-up Evaluation and Outcome Criteria Patients or their immediate relatives were contacted at 1, 3, and 6 months for the follow-up interviews. The information included hospitalization, readmission to ED, and mortality status. The mortality and ED readmissions of patients with and without frailty and sarcopenia were compared.

2.4 Statistical Analysis The data analysis was carried out using SPSS version 22. Kolmogorov-Smirnov test determined whether the numerical data were normally distributed. The numerical parameters exhibiting normal distributions were presented as mean (standard deviation), while those without normal distribution were shown as median (minimum-maximum). Non-quantitative parameters were analyzed using the Chi-square test and expressed as numbers and percentages. Student's t-test compared the numerical parameters with normal distribution between the groups, while the Mann-Whitney U test compared the non-parametric groups. Kruskal-Wallis and Bonferroni-adjusted Mann-Whitney U tests were conducted for the post hoc analysis. ANOVA and Tukey or Tamhane tests compared the means in more than two groups (according to the sarcopenia risk and frailty status). Spearman correlation test examined the relationship between numerical parameters. According to the Spearman test, the rho coefficient <0.4 was considered a weak correlation, 0.4 and 0.59 a moderate correlation, 0.6 and 0.79 a strong correlation, and 0.80 and above a very strong correlation. ROC analyses examined the potential of PRISMA-7 and SARC-F scores in predicting long-term mortality. The cut-off points were assessed using the ROC curve analysis. The best points for both scores (PRISMA-7 and SARC-F) were calculated using the Youden index. The significance level was considered as 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 65 years

Exclusion Criteria:

* Patients with no spontaneous heartbeat or breathing at the time of ED arrival

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged over 65 years and admitted to the emergency department
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Mortality | up to 6 months
Readmission to the Emergency Department | up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Firat University School of Medicine, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data will be available to the researchers, and they will be shared if wanted.